CLINICAL TRIAL: NCT01667120
Title: The Use of Ketorolac in Surgical Neonates
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-00554
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain Control in Surgical Neonates
Keywords: Ketorolac; postoperative pain; bleeding events
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Postoperative surgical neonates will receive an equivalent volume of 0.9% normal saline as placebo.
  Interventions: Drug: placebo
- Ketorolac (Experimental): Postoperative ketorolac 0.5mg/kg intravenously every 8 hrs for 72hrs will be administered.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Ketorolac 0.5mg/kg IV q8h x 72h.
  Other Names: Toradol
  Arms: Ketorolac
Drug: placebo — 0.9% normal saline 1ml/kg
  Other Names: 0.9% normal saline
  Arms: Placebo

SUMMARY:
The general purpose of this study is to characterize the safety profile of ketorolac in infants age 0-3 months. Our hypothesis is that ketorolac is safe in neonates, and effective in controlling pain with less narcotic administration required. Ketorolac 0.5mg/kg intravenously every 8 hrs for 72hrs will be administered versus an equivalent volume of 0.9% normal saline as placebo.

Primary: The primary purpose of this study is to compare bleeding events in neonates who receive ketorolac and those who do not receive ketorolac. The investigators hypothesize that ketorolac is safe and effective in infants > 37wks gestation and at least one week of age.

Secondary: The investigators intend to evaluate daily creatinine levels, pain scores, urine output per shift, platelet counts, hemoglobin levels, number of days on the ventilator, amount of narcotic administered, blood pressure, and reintubation events on all patients in this study as secondary study points.

DETAILED DESCRIPTION:
This is a Phase II, single center, randomized controlled pilot study. Hospitalized patients one week of age to 3 months of age who undergo an abdominal surgical procedure within the moderate or severe degree of pain category (see attached Table 1: postoperative pain categories) will be randomized to receive standard pain management regimens plus placebo (0.9% saline of equivalent volume) or ketorolac 0.5mg IV q8h x 72h plus standard pain management regimens. The postoperative management will be unchanged and at the discretion of the attending surgeon, as appropriate for the surgical procedure. The patients will be followed for 5 days, or 48hrs from the end of ketorolac therapy for primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Infants gestational age > 37 weeks and greater than or equal to one week of age to 3 months of age
2. Infants who are undergoing a surgical procedure on the abdomen
3. the parent or guardian has given informed consent.

Exclusion Criteria:

1. Gestational age < 37 weeks
2. Age less than one week or greater than 3 months of age
3. Known renal disease/dysplastic kidneys
4. Serum Creatinine > 0.4
5. Patients who have rising creatinine levels the day prior to surgery (increase of at least 1.5-fold from baseline)
6. Patients who are currently receiving other potentially renal toxic drugs or drugs that may interfere with hemostatic pathways as part of their clinical care (including but not limited to furosemide, hydrochlorothiazide, vancomycin, gentamicin, aspirin, tpa [except for use of thrombosed central venous catheters], enalapril, systemic heparin [except for use in central venous catheter flushes])
7. Patients who undergo nephrectomy
8. Patients with necrotizing enterocolitis
9. Patients with a hemoglobin value < 10g/dL
10. Recent (within 3 months) GI bleeding, ulceration, and/or perforation
11. Platelet count < 50,000
12. Ongoing disseminated intravascular coagulation or history of intraventricular hemorrhage
13. Recent (within 2 weeks) use or current use of other nonsteroidal anti-inflammatory drugs (NSAIDS) besides aspirin (ASA)
14. Allergy to ASA or other NSAIDS

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-07 (Estimated); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Safety from bleeding events. | 5 days
  Primary: The primary purpose of this study is to compare bleeding events in neonates who receive ketorolac and those who do not receive ketorolac. We hypothesize that ketorolac is safe and effective in infants > 37wks gestation and at least one week of age.

SECONDARY OUTCOMES:
Clinical parameters related to pain. | 5 days
  We intend to evaluate daily creatinine levels, pain scores, urine output per shift, platelet counts, hemoglobin levels, number of days on the ventilator, amount of narcotic administered, blood pressure, and reintubation events on all patients in this study as secondary study points.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Aldrink, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2013-01-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT01667120/Prot_000.pdf